CLINICAL TRIAL: NCT07186842
Title: First-in-human, Open-label, Multi-site, Phase I/IIa, Dose Escalation Trial With Expansion Cohorts to Evaluate Safety and Preliminary Efficacy of BNT329 in Participants With Advanced Solid Tumors Known to Express CA19-9
Brief Title: A Clinical Trial to Test if the Investigational Drug BNT329 is Safe and Potentially Beneficial for People With Advanced Solid Tumors Known to Express the Tumor Marker CA19-9
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT329-01; 2025-522613-26-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Cancers
Keywords: CA19-9; Anti-drug conjugate (ADC); Pancreatic ductal adenocarcinoma; Bile duct cancer; Colorectal cancer; Gastroesophageal junction cancer; Endometrial cancer; Ovarian cancer; Invasive urothelial carcinoma of the bladder and urinary tract
MeSH Terms: conditions — Bile Duct Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation - Part A (Experimental): BNT329 administered once every 3 weeks at protocol-defined dose levels
  Interventions: Drug: BNT329
- Dose Escalation - Part B (Experimental): BNT329 administered once every 2 weeks at protocol-defined dose levels
  Interventions: Drug: BNT329
- Dose Escalation: Part C (Experimental): BNT329 administered after pre-dosing with a CA19-9 targeting monoclonal antibody
  Interventions: Drug: BNT329; Drug: CA19-9-targeting monoclonal antibody
- Dose Expansion - Part D (Experimental): Participants will be randomized to one of two arms evaluating two different doses as selected from Parts A, B, and C
  Interventions: Drug: BNT329

INTERVENTIONS:
Drug: BNT329 — Intravenous (IV) infusion
Drug: CA19-9-targeting monoclonal antibody — Monoclonal antibody
  Arms: Dose Escalation: Part C

SUMMARY:
The main goal of this study is to evaluate the safety of BNT329 and to identify the best dose of BNT329. This will be done by measuring the number of side effects that participants experience and how severe they are.

The second goal of this study is to evaluate how well BNT329 works. This will be done by measuring the number of participants who respond to the treatment. The length of time where the tumor does not grow or spread will also be measured.

The study will also evaluate how BNT329 moves into, through, and out of the body and how the treatment affects the body.

DETAILED DESCRIPTION:
The study will consist of up to four parts (Parts A, B, C, and D).

Parts A, B, and C will be a dose escalation to investigate the safety and tolerability of BNT329. Parts A, B, and C will enroll participants with the following advanced solid tumors known to express carbohydrate antigen 19-9 (CA19-9): pancreatic ductal adenocarcinoma (PDAC) (the most common type of pancreatic cancer), bile duct cancer, a certain type of bladder cancer that started in the lining of the bladder or urinary tract (invasive urothelial carcinoma of the bladder and urinary tract), colorectal cancer, gastroesophageal junction cancer, endometrial cancer, or ovarian cancer. The cancer must not have responded well to previous treatments.

The study will start with recruitment into Part A. Part B (testing a more frequent dosing schedule) and Part C (testing pre-dosing with a CA19-9 targeting monoclonal antibody prior to BNT329 administration) will only be opened if indicated by cumulative data from the study.

Part D will be a dose optimization and proof-of-concept study to further investigate the safety and tolerability of BNT329 and to investigate preliminary anti-tumor activity. Part D will enroll participants with second-line plus PDAC.

Parts A, B, and C will be non-randomized. In Part D, participants will be randomized (1:1) into one of two arms which will evaluate two dose levels (as selected from Parts A, B, and C).

The study consists of a screening period, a treatment period, an End of Treatment Visit, two Safety Follow-Up Visits, and a survival follow-up period. The treatment period will last for a maximum of 2 years. Participants will remain in the survival follow-up until death, withdrawal of participant's consent, or termination of the study, whichever occurs first.

ELIGIBILITY:
Key Inclusion Criteria

All participants and parts:

* Have an ECOG PS of 0 to 1
* Have measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1), except for ovarian cancer where participants will be evaluated according to Gynecologic Cancer InterGroup criteria.
* Have a life expectancy of ≥3 months in the opinion of the investigator.
* Have adequate organ, coagulation, and hematologic function as defined in the protocol.

Parts A, B, and C:

* Have a histologically confirmed advanced/metastatic tumor type that is known to express CA19-9: PDAC, carcinoma of the bile ducts, invasive urothelial carcinoma of the bladder and urinary tract, colorectal adenocarcinoma, adenocarcinoma of the esophagogastric junction, endometrial carcinoma, and epithelial ovarian cancer (including adenocarcinoma of the fallopian tube and peritoneal epithelial cancer [except mesothelioma]).
* Have no available standard of care therapy likely to confer clinical benefit in the opinion of the investigator. Participants must have received all available standard therapies, including targeted therapies based on mutation status (per guidelines from the Food and Drug Administration, American Society of Clinical Oncology, European Society for Medical Oncology, or local guidelines used at the site), and failed at least first-line standard of care therapy prior to enrollment.

Part D:

* Have a histologically confirmed diagnosis of PDAC.
* Have received at least one prior systemic treatment regimen for advanced/metastatic disease. Participants who have progressed on <6 months of (neo)adjuvant chemotherapy can be included in the study.
* Have radiographic disease progression and no available standard of care therapy likely to confer clinical benefit in the opinion of the investigator.

Key Exclusion Criteria

All participants and parts:

* Are enrolled in another investigational study or are subject to exclusion periods from another investigational study.
* Have had an inadequate washout period for prior anticancer treatment prior to the first dose of investigational medicinal product (IMP) as defined in the protocol.
* Have received systemic steroids (>10 mg/day of prednisone or its equivalent) or other immunosuppressive therapy within 2 weeks prior to the first dose of IMP. The following are exceptions to this criterion:

  * Inhaled sprays, topical steroids, or local steroid injections (e.g., intra-articular injection).
  * Systemic steroids at physiological doses as replacement therapy (e.g., physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency).
  * Steroids as pre-medication for hypersensitivity reactions (e.g., computed tomography (CT) scan pre-medication).
* Have received any live vaccine within 4 weeks prior to the first dose of IMP or intend to receive a live vaccine during the study.
* Have brain metastases or spinal cord compression unless asymptomatic or treated and stable off steroids and anticonvulsants for at least 2 weeks prior to the first dose of IMP.
* Have a history of (noninfectious) interstitial lung disease (ILD)/pneumonitis that requires steroids, current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Have active gastric and duodenal ulcers, ulcerative colitis, or other gastrointestinal conditions that may cause bleeding or perforation in the opinion of the treating investigator.
* Have an active infection that requires systemic therapy within 1 week prior to the first dose of IMP. Participants receiving prophylactic anti-infective therapy (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) may be eligible after discussion with the sponsor.
* Have unresolved toxicities from previous anticancer therapy as defined in the protocol.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Parts A, B, and C - Occurrence of dose-limiting toxicities within a participant | First 21 days (Part A) or 28 days (Part B) after the first dose of BNT329.
  Per dose level/cohort.
All parts - Occurrence of treatment-emergent adverse events (TEAEs), Grade ≥3 TEAEs, serious adverse events (SAEs), treatment-related TEAEs, treatment-related Grade ≥3 TEAEs, and treatment-related SAEs | From first dose of BNT329 until 60 days after the last dose of BNT329 (up to 26 months).
  Per dose level/cohort/arm.
All parts - Occurrence of dose interruptions, reductions, and discontinuation of BNT329 due to TEAEs | From the time of initiation of the first dose of BNT329 until 60 days after the last dose of BNT329 (up to 26 months).
  Per dose level/cohort/arm.
Part D - Objective response rate (ORR) | From first dose of BNT329 until end of study (up to approximately 36 months).
  Per dose level/arm. Defined as the proportion of participants in whom a confirmed complete response (CR) or partial response (PR) (based on the investigator's assessment) is observed as best overall response.

SECONDARY OUTCOMES:
All parts - Assessment of area under the curve derived from serum concentrations of CA19-9-unbound ADC, CA19-9-unbound total anti-CA19-9 antibody, and unconjugated YL0010014 payload | First 21 days (Part A) or 28 days (Part B) after the first dose of BNT329.
  Per dose level/cohort/arm (if data permit)
All parts - Assessment of maximum concentration derived from serum concentrations of CA19-9-unbound ADC, CA19-9-unbound total anti-CA19 antibody, and unconjugated YL0010014 payload | First 21 days (Part A) or 28 days (Part B) after the first dose of BNT329.
  Per dose level/cohort/arm (if data permit).
All parts - Assessment of time to reach maximum concentration derived from serum concentrations of CA19-9-unbound ADC, CA19-9-unbound total anti-CA19-9 antibody, and unconjugated YL0010014 payload | First 21 days (Part A) or 28 days (Part B) after the first dose of BNT329.
  Per dose level/cohort/arm (if data permit).
All parts - Assessment of terminal half-life derived from serum concentrations of CA19-9-unbound ADC, CA19-9-unbound total anti-CA19-9 antibody, and unconjugated YL0010014 payload | First 21 days (Part A) or 28 days (Part B) after the first dose of BNT329.
  Per dose level/cohort/arm (if data permit).
Parts A, B, and C - ORR | From first dose of BNT329 until end of study (up to approximately 36 months).
  Per dose level/cohort. Defined as the proportion of participants in whom a confirmed CR or PR (based on the investigator's assessment) is observed as best overall response.
All parts - Disease control rate | From first dose of BNT329 until end of study (up to approximately 36 months).
  Per dose level/cohort/arm. Defined as the proportion of participants in whom a CR or PR or stable disease (assessed at least 6 weeks [±2 days] after the first BNT329 dose) is observed as best ORR per investigator's assessment.
All parts - Duration of response | From first dose of BNT329 until end of study (up to approximately 36 months).
  Per dose level/cohort/arm. Defined as the time from first objective response (CR or PR) to first occurrence of objective tumor progression (PD) or death from any cause, whichever occurs first.
All parts: Anti-drug antibody (ADA) prevalence | From first dose of BNT329 until up to 60 days after the last dose of BNT329 (up to 26 months).
  Per dose level/cohort/arm. Defined as the proportion of participants who are ADA positive at any timepoint (either baseline or post-baseline) (if data permit).
All parts - ADA incidence | From first dose of BNT329 until up to 60 days after the last dose of BNT329 (up to 26 months).
  Per dose level/cohort/arm. Defined as the proportion of participants having treatment-emergent ADA (if data permit).

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Response Person, Study Director — BioNTech SE
Locations (1):
- Florida Cancer Specialists, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No